CLINICAL TRIAL: NCT00752947
Title: Multi-Centre, Prospective, Open Label, Randomized Trial to Assess the Efficacy and Safety of Moxifloxacin Versus Levofloxacin Plus Metronidazole in the Treatment of Community-Acquired Pneumonia With Aspiration Factors
Brief Title: Efficacy and Safety Trial to Assess Moxifloxacin in Treating Community-Acquired Pneumonia (CAP) With Aspiration Factors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Prof. Sun Tieying, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOHBJH-STY-1
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Community-Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Moxifloxacin; Levofloxacin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: moxifloxacin
- B (Active Comparator)
  Interventions: Drug: levofloxacin; Drug: metronidazole

INTERVENTIONS:
Drug: moxifloxacin — Moxifloxacin 400mg iv. OD followed by moxifloxacin 400mg OD orally, 2-4 weeks.
  Other Names: Avelox
  Arms: A
Drug: levofloxacin — Levofloxacin 400mg i.v. OD followed by oral levofloxacin 400mg OD, 2-4 weeks
  Arms: B
Drug: metronidazole — metronidazole 0.5g i.v. bid followed by oral metronidazole 0.2g tid, 2-4 weeks
  Arms: B

SUMMARY:
The purpose of this study is to determine whether moxifloxacin in comparison to levofloxacin plus metronidazole are effective and safe in the treatment of community-acquired pneumonia with aspiration factors.

DETAILED DESCRIPTION:
186 patients in 4 centers will be enrolled in this study. Patients accord with the criteria of CAP with aspiration factors will be enrolled and randomized to one of the following groups. The treatment duration will range from 2 to 4 weeks.

Study Group: Intravenous treatment with moxifloxacin 400mg i.v. OD. Based on investigator's decision, a switch can be made to moxifloxacin 400 mg OD, orally (Moxifloxacin injection will be used no more than 3 weeks consecutively) .

Control Group: Intravenous treatment with levofloxacin 400mg i.v. OD plus metronidazole 0.5g i.v. bid. Based on investigator's decision, a switch can be made to levofloxacin 400mg OD plus metronidazole 0.2g tid, orally.

Treatment should be continued until complete resolution of the radiological, clinical and laboratory alterations or until no further regression can be observed. Clinical, bacteriological, laboratory and radiological examinations will be performed pre-treatment. Swallowing/coughing reflection test will be used for aspiration factor diagnosis. Risk factors (Decreased level of consciousness, dysphagia, gastroesophageal reflux, neurologic disease, mechanical and device-related (e.g. nasogastric feeding tube) impairment of upper aerodigestive tract, vomiting, bronchial obstruction due to neoplasm or foreign body, bronchiectasis, pulmonary infarction, etc) will be evaluated before the treatment. Clinical and laboratory examinations such as blood routine(including Hb, differential blood count, etc), urine routine, biochemistry examination (including serum bilirubin, hepatic/renal function parameters, etc), coagulation examination will be repeated selectively. Radiological examination (e.g. chest x-ray) will be repeated at each visit for clinical monitoring after one week treatment. At the test-of-cure visit (7-14 days after the end of therapy) comprehensive clinical, bacteriological and laboratory examinations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or above.
* Patients who are willing and able to provide written informed consent.
* Accord with the diagnosis criteria of CAP based on clinical, radiological and microbiological findings.
* With aspiration factors (Including swallowing or coughing reflection test positive)

Exclusion Criteria:

* Known hypersensitivity to fluoroquinolones and/or metronidazole.
* Female patients who are pregnant or lactating.
* Patients with mechanical ventilation lasting more than 48 hours prior to enrollment.
* Patients with neutropenia (neutrophil count <1.000/mm3) due to malignancy or chemotherapy.
* Patients with a severe, life-threatening disease with a life expectancy of less than 2 months.
* Patients with a co-existent disease considered likely to affect the outcome of the study (e.g. lung cancer, cystic fibrosis, collagen vascular disease affecting the lungs, pleural empyema, severe cardiac failure class III or IV of the NYHA).
* Patients with poststenotic pneumonia (e.g. in connection with carcinoma of the lung).
* Patients with acute infarction pneumonia.
* Patients with active pulmonary tuberculosis.
* Patients with lung abscess/pneumonia with concomitant endocarditis.
* Patients with known i.v. drug abuse.
* Patients known to have AIDS (CD4 count <200/ul) or HIV-seropositives who are receiving HAART (highly activated antiretroviral therapy). Note: HIV-positive patients may be included. HIV testing is not required for this study protocol.
* Patients with severe hepatic impairment (Child-Pugh C).
* Patients on hemodialysis, equivalent to creatinine clearance <15 ml/min/1.73 m2.
* Patients known to have congenital or sporadic syndromes of QTc prolongation, or are receiving concomitant medication reported to increase the QTc interval, e.g. amiodaron, sotalol, disopyramide, quinidine, procainamide, terfenadine.
* Previous history of tendinopathy with quinolones.
* Patients who have previously been included in this study.
* Patients with any investigational drug within 30 days of screening.
* Patients requiring concomitant systemic antibacterial agents.
* Pre-treatment with a systemic antibacterial agent within 24 hours prior to enrollment (Except for the cases that pre-treatment is not effective based on the clinical judgment).
* Severe CAP.
* Other contraindications in package insert.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Test-of-cure visit (7-14 days after the end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Tieying Sun, Principal Investigator — Beijing Hospital
Locations (2):
- China (2):
  - Tieying Sun, Beijing
  - Xiuhong Nie, Beijing